CLINICAL TRIAL: NCT03564535
Title: Comparison of Mesh Fixation With Tackers to Use of Self Fixating Mesh in Total Extra Peritoneal Inguinal Hernia Repair: A Double Blinded Randomized Controlled Trial
Brief Title: Comparison of Self Fixating Mesh to Mesh Fixation With Metallic Tacks in Laparoscopic Inguinal Hernia Repair
Acronym: SELFITAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Tushar Subhadarshan Mishra, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T/IM-NF/Surg/17/36
Record Dates: First submitted 2018-04-10; First posted 2018-06-21 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Inguinal Hernia; Adult
Keywords: Adult; Inguinal hernia; Inflammatory; Surgical Mesh; Laparoscopy/Methods; Postoperative pain; Recurrence; Randomized Controlled Trials; Double-Blind Method; Pain; Chronic pain; Seroma; Total extraperitoneal repair; Tacker; Mesh fixation; Self gripping
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Recurrence; Pain; Chronic Pain; Seroma

STUDY DESIGN:
Intervention Model Description: Patients of uncomplicated inguinal hernia presenting to the outpatient department of AIIMS, Bhubaneswar will be recruited to the study. They would be put either in the conventional tacker group or self-fixating mesh group based on the sealed envelope which will be revealed once the patient is intubated. Random allocation done using random allocation software. Surgeries would be performed by single surgery team experienced in laparoscopic hernia repair.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and follow-up clinician will be blinded regarding the use of mesh fixation. The mesh fixation technique will only be entered in the master chart of the student but not in the Operation notes, in order to prevent accidental disclosure by a curious patient or follow up evaluator instead the phrase, "TEP done by 11x15cm mesh will be written.'' For legal reasons details of the tack applicator device will be recorded on the nursing count sheet.) Follow-up will be performed by a different clinician to the operating surgeon. There would be no external clues such as differences in the location or size of skin incisions to indicate whether fixation had been performed or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SELF FIXATING GROUP (Experimental): Monofilament polyester mesh with polylactic acid (PLA) microgrips of size 11*15 will be used. It is an isoelastic large-pore knitted fabric with a density of 73g/m2 at implantation and 38g/m2 after microgrips absorption which will be at 18 months. The resorbable micro grips provide immediate adherence to surrounding muscle and adipose tissue during the initial days post hernia surgery, serving as an alternate method of fixation to traditional sutures, tacks, staples, or fibrin sealants. No additional tacks, staples, sutures, or fibrin sealant will be used.
  Interventions: Device: Self fixating group
- TACKER FIXATION GROUP (Active Comparator): Patients will be undergoing mesh ﬁxation with non-absorbable tacks. The tacks would be used such that they avoid bony prominences and vascular and neural structures. One or two tacks will be put at the Cooper's ligament and another applied laterally superior to the iliopubic tract in the anterior abdominal wall. In any patient, the maximum number of tacks applied will not exceed three.
  Interventions: Device: Tacker fixation group

INTERVENTIONS:
Device: Self fixating group — Monofilament polyester mesh with polylactic acid (PLA) microgrips of size 11*15 will be used. It is an isoelastic large-pore knitted fabric with a density of 73g/m2 at implantation and 38g/m2 after microgrips absorption which will be at 18 months. The resorbable micro grips provide immediate adherence to surrounding muscle and adipose tissue during the initial days post hernia surgery, serving as an alternate method of fixation to traditional sutures, tacks, staples, or fibrin sealants. No additional tacks, staples, sutures, or fibrin sealant will be used.
  Other Names: Monofilament polyester mesh with polylactic acid microgrips
  Arms: SELF FIXATING GROUP
Device: Tacker fixation group — Patients will be undergoing polyester mesh ﬁxation with non-absorbable tacks. The tacks would be used such that they avoid bony prominences and vascular and neural structures. One or two tacks will be put at the Cooper's ligament and another applied laterally superior to the iliopubic tract in the anterior abdominal wall. In any patient, the maximum number of tacks applied will not exceed three.
  Other Names: Polyester mesh with tack fixation
  Arms: TACKER FIXATION GROUP

SUMMARY:
This study compares the use of self-fixating mesh to mesh fixation with tackers in the management of inguinal hernia by laparoscopic method. Half of the participants in the study will be treated using self-fixating mesh, while the other half will be treated using conventional mesh fixed with tackers.

DETAILED DESCRIPTION:
Conventional tacker mesh fixation group Patients will be undergoing mesh ﬁxation with non-absorbable tacks. Monofilament polyester mesh of size 15*11cm will be used. The tacks would be used such that they avoid bony prominences and vascular and neural structures. One tack will put at the Cooper's ligament and another applied laterally superior to the iliopubic tract in the anterior abdominal wall. In any patient, the maximum number of tacks applied will not exceed four. Preperitoneal space will be deﬂated under direct visualization after the mesh is placed. Hernia sac and any cord lipoma will be placed behind the mesh. During the deﬂation process, repositioning of the peritoneal sac on the mesh, in particular the dorsal edge of the latter would be carefully performed to avoid displacement or folding of the mesh.

Self-fixating mesh group In this group,Monofilament polyester mesh with polylactic acid (PLA) microgrips of size 15*11 will be used. It is an isoelastic large-pore knitted fabric with a density of 73g/m2 at implantation and 38g/m2 after microgrips absorption which will be at 18 months. The resorbable micro grips provide immediate adherence to surrounding muscle and adipose tissue during the initial days post hernia surgery, serving as an alternate method of fixation to traditional sutures, tacks, staples, or fibrin sealants. No additional tacks, staples, sutures, or fibrin sealant is used

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral inguinal hernia
2. Age 18-80years
3. American Society of Anesthesiologists (ASA) Grade 1 or 2

Exclusion Criteria:

1. Patient unfit for general anesthesia or laparoscopic surgery
2. Large scrotal hernias
3. Irreducible hernias
4. Morbid obesity
5. Previous pelvic surgery
6. Coagulopathy
7. Those who cannot understand the VAS score
8. Those who did not agree to participate in the study
9. Gastritis
10. Gastroesophageal reflux disease
11. Liver dysfunction
12. kidney dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in post operative pain | 1 hour, 6 hours,12 hours, 24 hours, 7 days, 1 month and 3 months post surgery
  Postoperative pain will be evaluated using Visual Analogue Scale (0 TO 10) at follow up at ward, Out Patient Department/patient's pain diary/by telephonic call/by e-mail. In the first 6hours, if the VAS score >4 Inj.Paracetamol 1gm I V will be given, if the VAS score >4 after 30min of previous dose, inj diclofenac 75mg iv will be given, if VAS score is still >4 inj.Tramadol 100mg will be given. After 6 hours pain killers will be given in the same order and same dose orally as a tablet depending upon the requirement and pain score. Highest pain score at any given point of time and average pain score will be calculated.

SECONDARY OUTCOMES:
Mesh displacement | 24 hours and 1 month post surgery
  Meshes will be marked with three 5-mm surgical clips at its medial inferior, medial superior and lateral inferior corners. Pelvic x ray will be done on post operative day 1 and at the end of 1 month to look for any displacement.
Inflammatory markers | On the day of surgery (pre op), 48 hours post surgery, 3 months post surgery
  On the day of surgery, preoperative venous blood samples (baseline) will be withdrawn and assayed for C-reactive protein (CRP) levels, erythrocyte sedimentation rate (ESR), and total white blood cell count (WBC). Venous blood samples will be obtained 48 h post-surgery and assayed for CRP and WBC. ESR will be checked at 3 months postoperatively. Acute surgical trauma corresponding to postoperative acute pain will be measured using CRP and WBC, while chronic pain will be measured with ESR.
Post operative complications | 6 hours, 24 hours, 48 hours, 7 days, 1 month, 3 months post surgery
  Various known post operative complications will be looked for such as
  1. Post-operative urinary retention
  2. Seroma
  3. Hematoma
  4. Early recurrence
  5. Wound infection
  6. Cord edema
  7. Testicular atrophy
Operative time | Time of skin incision to time of skin closure
  Time required to complete the surgery i.e from incision time to closure time.
Achieving criteria of fitness for discharge | Time of skin closure to time of discharge which will be approximately 2 days.
  Discharge criteria includes
  1. Pain adequately controlled by oral analgesics (VAS Score <4)
  2. Ambulation without help
  3. Absence of post operative complications requiring surgical interventions
Resumption to normal activities | Immediate post operative period.
  Return to normal activity will be assessed by recording the time taken by the patient to get in and out of bed and ambulate without help.
Total cost towards the mesh and its fixation | Immediate post operative period.
  Total cost involved in the procedure would be measured in both the arms.
Quality of life using Carolinas Comfort Scale | 6 hours, 24 hours, day 7 , 1 month and 3 month post surgery.
  Quality of life will be measured using Carolinas Comfort Scale (CCS), a validated post hernia quality of life and pain assessment tool developed by physician and researchers from Carolina laparoscopic and advanced surgery programme (CLASP), to monitor quality of life in patients undergoing hernia repair. The CCS is a 23-item, Likert type questionnaire that measures, on a scale of 0 to 5, severity of pain, sensation and movement limitations from the mesh.
  Carolinas Comfort Scale questionnaire (maximum: 115 points)
  Sensation of mesh, pain and movement limitations need to be graded on a scale of 0 to 5 or as not applicable
  1. While laying down,
  2. While bending over,
  3. While sitting up, 4.While performing activities of daily living (getting out of bed, bathing, getting dressed),
  5 When coughing or deep breathing, 6 When walking or standing, 7 When walking up or down stairs, 8 When exercising (other than work-related), Total CCS score: ………
Mesh deployment time | Time from insertion of mesh into trocar till complete deployment is done.
  Total time required from insertion of mesh into trocar till complete deployment is done. Mesh deployment satisfaction rate will also be noted.
Intra operative complications | Intra operatively
  Various intra operative complications will be recorded such as
  1. Bladder injury
  2. Vas Deferens injury
  3. Iliac vein injury
  4. Pneumoperitoneum
  5. Dropping down/Injury of inferior epigastric artery
  6. Bowel injury

CONTACTS AND LOCATIONS:
Locations (1):
- Tushar S Mishra, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liew W, Wai YY, Kosai NR, Gendeh HS. Tackers versus glue mesh fixation: an objective assessment of postoperative acute and chronic pain using inflammatory markers. Hernia. 2017 Aug;21(4):549-554. doi: 10.1007/s10029-017-1611-1. Epub 2017 Apr 17. PMID 28417279
- [Result] Buyukasik K, Ari A, Akce B, Tatar C, Segmen O, Bektas H. Comparison of mesh fixation and non-fixation in laparoscopic totally extraperitoneal inguinal hernia repair. Hernia. 2017 Aug;21(4):543-548. doi: 10.1007/s10029-017-1590-2. Epub 2017 Feb 18. PMID 28214943
- [Result] Garg P, Rajagopal M, Varghese V, Ismail M. Laparoscopic total extraperitoneal inguinal hernia repair with nonfixation of the mesh for 1,692 hernias. Surg Endosc. 2009 Jun;23(6):1241-5. doi: 10.1007/s00464-008-0137-0. Epub 2008 Sep 24. PMID 18813990
- [Result] Bresnahan E, Bates A, Wu A, Reiner M, Jacob B. The use of self-gripping (Progrip) mesh during laparoscopic total extraperitoneal (TEP) inguinal hernia repair: a prospective feasibility and long-term outcomes study. Surg Endosc. 2015 Sep;29(9):2690-6. doi: 10.1007/s00464-014-3991-y. Epub 2014 Dec 18. PMID 25519425
- [Result] Teng YJ, Pan SM, Liu YL, Yang KH, Zhang YC, Tian JH, Han JX. A meta-analysis of randomized controlled trials of fixation versus nonfixation of mesh in laparoscopic total extraperitoneal inguinal hernia repair. Surg Endosc. 2011 Sep;25(9):2849-58. doi: 10.1007/s00464-011-1668-3. Epub 2011 Apr 13. PMID 21487873